CLINICAL TRIAL: NCT03397459
Title: Cervicobrachial Neuralgia and Sagital Balance of the Cervical Spine
Acronym: CNSBS-NCBES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/284
Record Dates: First submitted 2017-12-21; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Cervicobrachial Neuralgia; Lordosis
Keywords: cervicobrachial neuralgia; sagittal balance; lordosis
MeSH Terms: conditions — Brachial Plexus Neuritis; Lordosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spine teleradiography EOS

SUMMARY:
The aim of this observational study is to establish estimation of global lordosis of the cervical spine (from C3 to C7) in patients with cervicobrachial neuralgia.

DETAILED DESCRIPTION:
The main judgement critearia is the estimation in degree of this lordosis measured on EOS radiographies, The study includes adults patients with non traumatic cervicobrachial neuralgia caused by discal hernia free from any previous spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old)
* Suffering of cervicobrachial neuralgia caused by cervical hernia on MRI diagnosed by a neurosurgeon
* with social care rights

Exclusion Criteria:

* Post traumatic cervicobrachial neuralgia in the past 12 months
* Anteriority of spine surgery
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering of cervicobrachial neuralgia in the hospital of BESANCON, FRANCE followed by a neurosurgeon.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Low Cervical spine lordosis | Day 1
  In degree, the angle between the lower plate of C2 and the lower plate of the last cervical vertebrea (physiologycally)

SECONDARY OUTCOMES:
NDI | Day 1
  Pain questionnaires (score of 0 and 50)

CONTACTS AND LOCATIONS:
Locations (1):
- HAMDAN, Besançon, France

IPD SHARING:
Plan to Share IPD: No